CLINICAL TRIAL: NCT05934448
Title: A Phase II Trial of Pembrolizumab in Combination With Chimeric Antigen Receptor Therapy in Patients With Relapsed/Refractory Primary Mediastinal B-cell Lymphoma
Brief Title: Pembro Plus CAR T-cell Therapy in R/R in PMBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Crombie, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Crombie, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-179
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Primary Mediastinal Large B-cell Lymphoma (PMBCL); Primary Mediastinal Large B Cell Lymphoma; Primary Mediastinal Large B-Cell Lymphoma Refractory; Primary Mediastinal Large B-Cell Lymphoma Recurrent; Epstein-Barr Virus Positive Diffuse Large B-Cell Lymphoma; T-Cell/Histiocyte-Rich Large B-Cell Lymphoma
Keywords: Primary Mediastinal Large B-cell Lymphoma (PMBCL); Primary Mediastinal Large B Cell Lymphoma; Primary Mediastinal Large B-Cell Lymphoma Refractory; Primary Mediastinal Large B-Cell Lymphoma Recurrent; T-Cell/Histiocyte-Rich Large B-Cell Lymphoma; Epstein-Barr virus-positive diffuse large B-cell lymphoma
MeSH Terms: interventions — pembrolizumab; fludarabine; Cyclophosphamide; Receptors, Chimeric Antigen; Automobiles; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PEMBROLIZUMAB (Experimental): * Participants will undergo (leukapheresis) for manufacturing of commercial product as per standard of care (SOC) Cycle 1 Day -21or earlier
  * Pembrolizumab will be administered per protocol on cycle 1 day -20 and on day +1 following Chimeric Antigen Receptor (CAR) Therapy Infusion infusion, every 3 weeks for up to 2 years, unless there is confirmed progression of disease or unacceptable toxicity.
  * Upon the completion of successful manufacturing, patients will undergo lymphodepleting chemotherapy (fludarabine, cyclophosphamide) for chimeric antigen receptor (CAR) therapy infusion as per SOC.
  * Participants will receive Chimeric Antigen Receptor (CAR) Therapy Infusion (SOC) on day 0 in the hospital and will remain in the inpatient setting for observation for a minimum of 7 days or until CAR T-cell toxicities resolve to grade 1 or better. The choice of CAR-T product will be left to the discretion of the treating investigator.
  Interventions: Drug: Pembrolizumab; Drug: Lymphodepletion Chemotherapy; Drug: Chimeric Antigen Receptor (CAR) Therapy Infusion; Procedure: Leukapheresis

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab via iv, dosage and timing per protocol
  Other Names: Keytruda
Drug: Lymphodepletion Chemotherapy — Participants will undergo lymphodepleting chemotherapy (fludarabine, cyclophosphamide) for CAR T-cell therapy as per SOC
  Other Names: Fludarabine; Cyclophosphamide
Drug: Chimeric Antigen Receptor (CAR) Therapy Infusion — Day 0 in the hospital and will remain in the inpatient setting for observation for a minimum of 7 days or until CAR T-cell toxicities resolve to grade 1 or better. The choice of CAR-T product will be left to the discretion of the treating investigator.
Procedure: Leukapheresis — manufacturing using commercial product as per standard of care (SOC) Cycle 1 Day -21 or earlier

SUMMARY:
This research study is evaluating the combination of drugs, pembrolizumab with chimeric antigen receptor (CAR) T-cell therapy, as a possible treatment for primary mediastinal B-cell lymphoma that has recurred after prior treatment.

The names of the study drugs involved in this study are:

- Pembrolizumab

Standard treatment will include:

* CAR T-cell therapy (either axicabtagene-ciloleucel or lisocabtagene maraleucel)
* Cyclophosphamide
* Fludarabine

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The names of the study drugs involved in this study are:

- Pembrolizumab

Standard treatment will include:

* CAR T-cell therapy (either axicabtagene-ciloleucel or lisocabtagene maraleucel)
* Cyclophosphamide
* Fludarabine Participants will receive study treatment for up to 2 years and will be followed for 5 years. It is expected that about 35 people will take part in this research study.

The U.S. Food and Drug Administration (FDA) has approved pembrolizumab for this specific disease after two or more lines of therapy, but not in combination with CAR T-cell therapy.

The CAR T-cell therapies to be used in this study are axicabtagene-ciloleucel and lisocabtagene maraleucel. The U.S. FDA has approved axicabtageneciloleucel and lisocabtagene maraleucel as treatment options for this disease, but not in combination with pembrolizumab.

A small subset of patients with T-cell histiocyte-rich large B-cell lymphoma and EBV+ large B-cell lymphoma will also be included.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of PMBCL, EBV+ DLBCL or THRLBCL at one of the participating institutions.
* Availability of archival or freshly collected tumor tissue before study enrollment. If archival tissue is unavailable or is determined to be inadequate, tumor tissue must be obtained from a biopsy performed at screening, unless an exception is given after consultation with the sponsor-investigator.
* Eligible for standard of care CAR T-cell therapy with progression after at least two prior lines of therapy OR refractory to initial chemoimmunotherapy OR relapse within 12 months of front-line chemoimmunotherapy OR one prior line of therapy and not fit for HSCT.
* ECOG Performance Status of 0 or 1.
* Left ventricular ejection fraction (LVEF) ≥ 50% on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO).
* Adequate hematologic function (unless due to underlying disease, as established for example, by extensive bone marrow involvement or due to hypersplenism secondary to the involvement of the spleen by lymphoma per the investigator), defined as follows:

  * ANC ≥ 1,000/μL
  * Hemoglobin ≥ 8 g/dL
  * Platelet count ≥ 50,000/μL
* Participants must have adequate organ as defined below:

  * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
  * AST(SGOT)/ALT(SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver involvement)
  * Adequate renal function defined by serum creatinine ≤1.5 x ULN or creatinine clearance (by Cockcroft-Gault) ≥ 40 ml/min for patients with serum creatinine >1.5 x ULN
* At least one bi-dimensionally FDG-avid measurable lymphoma lesion on PET/CT scan, defined as ≥ 1.5 cm in its longest dimension on CT scan, or ≥ 1 cm if extranodal (and measurable).
* Women of childbearing potential (WOCBP) and men must agree to use effective contraception when sexually active. This applies for the time period between signing of the informed consent form and 6 months for WOCBP and for men after the last administration of study treatment. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for continuous 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control, e.g. intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner, use of two forms of birth control, and sexual abstinence. The use of condoms by male patients is required unless the female partner is permanently sterile.
* Age ≥18 years.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients in urgent need of cytoreductive therapy.
* Participants who are receiving any other investigational agents.
* History of other malignancies, except:

  * Malignancy treated medically or surgically with curative intent and with no known active disease present for ≥2 years before study registration
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease.
  * Localized prostate cancer and low-risk prostate cancer on active surveillance
  * In the opinion of the treating investigator, there is limited potential to interfere with the safety or efficacy of the investigational regimen. Such exceptions must be approved by the Sponsor-Investigator.
* Has received a live vaccine within 30 days prior to study registration. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Less than 6 months of response to prior PD-L1 inhibitor or PD-1 inhibitor or grade 3 or higher immune-related adverse events.
* Prior treatment with CAR T-cell therapy.
* Lactating or pregnant. Women of childbearing potential (WOCBP) must have a negative pregnancy test (urine or serum) at screening. WOCBP will require a negative pregnancy test within 72 hours prior to starting treatment, but eligibility for study enrollment may be confirmed based on testing at screening.
* Known active lymphomatous involvement of the central nervous system. History of prior CNS involvement is allowed.
* Recent infection requiring intravenous antibiotics that was completed ≤7 days before the first dose of study drug, or any uncontrolled active systemic infection.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus infection.
* History of Human immunodeficiency virus (HIV)-infection.
* Has received prior radiotherapy within 2 weeks of study registration. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has received prior systemic anti-cancer therapy within 2 weeks or investigational agents within 4 weeks.
* Significant liver disease, such as hepatitis (viral or non-viral) or cirrhosis
* Prior macrophage activation syndrome (MAS) or hemophagocytic lymphohistiocytosis (HLH)
* Uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months of enrollment.
* Known history of central nervous system or neurologic disease including stroke or intracranial hemorrhage within 3 months prior to enrollment or seizure disorder. Prior CNS involvement with lymphoma is allowed if previously treated with no evidence of involvement at study entry.
* Prior solid organ or allogeneic stem cell transplant or within 6 weeks of autologous stem cell transplant.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to study registration. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Active pneumonitis or interstitial lung disease.
* Severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has not met requirements for standard of care CAR-T therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2027-06-06 (Estimated); Study Completion 2031-06-06 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate at 6 Months | 6 months
  Per Lugano 2014 criteria, Complete Response (CR) is defined as PET-CT, score 1, 2, or 3* with or without a residual mass on 5 point scale; or on CT, target nodes/nodal masses must regress to ≤ 1.5 cm in LDi, and no extralymphatic sites of disease.

SECONDARY OUTCOMES:
Treatment-Related Grade 3 or Higher Cytokine Release Syndrome (CRS) Rate | 6 months
  CRS rate will be summarized based on American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading (Lee et al, 2019).
Treatment-Related Grade 3 or Higher Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) Rate | 6 months
  ICANS rate will be summarized based on ASTCT ICANS Consensus Grading for Adults using ICE 10-Point Neurological Assessment (Lee et al, 2019)
Treatment-Related Grade 3 or Higher Prolonged Cytopenia Rate | 6 months
  Prolonged cytopenias defined as Grade 3 or higher neutropenia, anemia, or thrombocytopenia persisting for ≥ 4 weeks from receiving CAR T-cell therapy based on CTCAEv5.
Treatment-Related Grade 3 or Higher Immune-Related Adverse Event (irAE) Rate | 6 months
  Composite rate comprised of all irAEs based on CTCAEv5
Complete Response (CR) Rate at 6 Months in patients with EBV+ DLBCL and THRLBCL | 6 months
  Per Lugano 2014 criteria, Complete Response (CR) is defined as PET-CT, score 1, 2, or 3* with or without a residual mass on 5 point scale; or on CT, target nodes/nodal masses must regress to ≤ 1.5 cm in LDi, and no extralymphatic sites of disease.
Partial Response (PR) Rate | baseline, 1 month, 3 month, and every 6 months up to 24 months
  Per Lugano 2014 criteria, partial response (PR) is defined as PET-CT Score 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size; or On CT ≥ 50% decrease in SPD of up to 6 target measurable nodes and extranodal sites; no increase in non-measured lesions; spleen if enlarged must have regressed by >50% in length beyond normal.
Duration of Response (DOR) | baseline, 1 month, 3 month, and every 6 months up to 24 months
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause. Participants without events reported are censored at the last disease evaluation). CR, PR and PD are defined based on Lugano 2014 criteria.
Median Progression-free survival (PFS) | Baseline, 1 month, 3 month (if not CR at 1 month) and then every 6 months until 24 months.
  Progression-Free Survival (PFS) based on Kaplan-Meier method is defined as the time from randomization (or registration) to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation. PD is defined based on Lugano 2014 criteria.
Median overall survival (OS) | Up to 5 years
  Overall Survival (OS) based on Kaplan-Meier is defined as the time from randomization (or registration) to death due to any cause or censored at date last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Crombie, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu